CLINICAL TRIAL: NCT06836778
Title: Comparative Study of Carvedilol Monotherapy Versus Combination Therapy With Endoscopic Variceal Ligation (EVL) for Primary Prophylaxis of Variceal Bleeding in Patients With Hepatocellular Carcinoma With High-Risk Esophageal Varices: A Randomized Trial
Brief Title: Comparative Study of Carvedilol Monotherapy Versus Combination Therapy With Endoscopic Variceal Ligation (EVL) for Primary Prophylaxis of Variceal Bleeding in Patients With Hepatocellular Carcinoma With High-Risk Esophageal Varices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HCC-08
Record Dates: First submitted 2025-01-27; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NSBB+EVL (Experimental): Non-selective beta blocker (Carvedilol 3.125 mg BD for 3 days followed by 6.25 mg BD , maximum dose would be 12.5 mg BD , same shall be switch to maximum tolerable dose if Systolic BP< 90 , H,R<55) + EVL every 3 weeks till eradication of varices followed by every 3 months
  Interventions: Drug: Carvedilol Tablets; Procedure: Endoscopic Variceal Ligation
- NSBB (Active Comparator): Non-selective beta blocker (Carvedilol 3.125 mg BD for 3 days followed by 6.25 mg BD , maximum dose would be 12.5 mg BD , same shall be switch to maximum tolerable dose if Systolic BP< 90 , H,R<55)
  Interventions: Drug: Carvedilol Tablets

INTERVENTIONS:
Drug: Carvedilol Tablets — Non-selective beta blocker (Carvedilol 3.125 mg BD for 3 days followed by 6.25 mg BD , maximum dose would be 12.5 mg BD , same shall be switch to maximum tolerable dose if Systolic BP< 90 , H,R<55)
Procedure: Endoscopic Variceal Ligation — EVL every 3 weeks till eradication of varices followed by every 3 months.
  Arms: NSBB+EVL

SUMMARY:
Esophageal varices are common in patients with hepatocellular carcinoma (HCC), with an incidence rate of 63% at the time of HCC diagnosis. Following an acute variceal bleed, the 6-week mortality rate for HCC patients is as high as 26%. Mortality rates escalate notably in HCC patients experiencing acute variceal bleeding, especially with increasing cancer severity indicated by BLCL status. Research suggests that the cumulative incidence rate of variceal bleeding at one year in patients receiving primary prophylaxis is almost half that of patients not receiving any prophylaxis.

Beta blockers are the standard therapy for primary prophylaxis in patients with portal hypertension to prevent variceal bleeding. Endoscopic band ligation has also shown promising results in recent studies. However, the combined impact of beta blockers and esophageal band ligation on lowering the incidence of variceal bleeding remains unstudied.

The aim of this study is to compare the efficacy of carvedilol monotherapy versus combination therapy with carvedilol and endoscopic band ligation in patients with HCC for primary prophylaxis of high-risk esophageal varices.

DETAILED DESCRIPTION:
Study population: All patients aged ≥ 18 years and ≤ 80 years admitted in Institute of Liver and Biliary Sciences, New Delhi with HCC of any cause and high risk esophageal varices and are giving written consent for participation in the study.

Study design - Single center, Open label, Randomized controlled trial Study period - 6 months Intervention - The patients will be randomized into Group -A (NSBB arm) and Group-B (EVL + NSBB arm). Both the group will receive the remaining treatment as per protocol Group A: Non-selective beta blocker (Carvedilol 3.125 mg BD for 3 days followed by 6.25 mg BD , maximum dose would be 12.5 mg BD , same shall be switch to maximum tolerable dose if SBP< 90 , H,R<55) Group B: Non-selective beta blocker (Carvedilol 3.125 mg BD for 3 days followed by 6.25 mg BD , maximum dose would be 12.5 mg BD , same shall be switch to maximum tolerable dose if SBP< 90 , H,R<55) + EVL every 3 weeks till eradication of varices followed by every 3 months.

Monitoring and assessment: Monitoring and evaluation would be done once a month for first 3 months then at 6th month.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Cirrhosis with HCC
3. High risk oesophageal varices (*large or small with RCS)
4. Valid consent

Exclusion Criteria:

1. Any contra-indication to beta-blockers
2. Any EVL or Sclerotherapy within last 3 months
3. Any past history of TIPS or surgery for portal hypertension
4. HCC with BCLC-D
5. Patients with past history of variceal bleed.
6. Patient With Liver transplant expected in next 2 weeks would be excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients of cirrhosis with HCC and high risk oesophageal varices on carvedilol developing variceal bleed with or without EVL in 6months follow up. | 6 months

SECONDARY OUTCOMES:
Proportion of patient developing variceal bleed while on therapy with Tyrosine Kinase Inhibitors despite on carvedilol with or without EVL | 6 months
Proportion of patient developing variceal bleed while on therapy with immunotherapy despite on carvedilol with or without EVL. | 6 months
Percentage of patient of cirrhosis with HCC and Portal Vein Tumoral Thrombosis developing variceal bleed while on carvedilol with or without EVL. | 6 months
Proportion of patients having post-EVL ulcer bleed after endoscopic variceal ligation. | 6 months
Proportion of patients with change in non invasive test for portal hypertension in both groups. | 6 months
  Non invasive markers: LSM, SSM, APRI Score, ALBI Score
Proportion of patient developing variceal bleed after SBRT for advanced Hepatocellular carcinoma | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided